CLINICAL TRIAL: NCT00021736
Title: Phase II/III Randomized, Double-Masked, Trial, to Establish the Safety and Efficacy of Intravitreal Injections of EYE001 (Anti-VEGF Pegylated Aptamer) Given Every 6 Weeks for 54 Weeks, in Patients With Exudative AMD).
Brief Title: Phase II/III Study of Anti-VEGF in Neovascular AMD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eyetech Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EOP1004B
Record Dates: First submitted 2001-08-03; First posted 2001-08-06 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-07

CONDITIONS: Macular Degeneration; Choroidal Neovascularization
Keywords: choroidal neovascularization (CNV); subretinal neovascularization
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization

INTERVENTIONS:
Drug: EYE001 anti-VEGF aptamer

SUMMARY:
The purpose of the study is to determine whether the anti-VEGF drug is effective at stabilizing and/or improving vision in patients with the wet form of AMD

DETAILED DESCRIPTION:
This will be a randomized, double-masked, controlled, dose-ranging, multi-center comparative trial, in parallel groups. Patients will be stratified by clinical center, by percentage of classic CNV vessels: [predominantly classic (>50%) vs. minimally classic (1-49%) vs. purely occult (0%)], and according to whether, or not, they have received prior PDT with Visudyne (no more than once). All patients will be re-randomized after 54 weeks of treatment to either, continue or discontinue therapy for further 48 weeks.

ELIGIBILITY:
Patients of either gender, aged 50 years or above, diagnosed with subfoveal CNV secondary to AMD and with best corrected visual acuity of 20/40 to 20/320 in the absence of subfoveal atrophy or scarring in the study eye, and better or equal to 20/800 in the fellow eye, may be enrolled. Clinically significant concomitant diseases will be excluded.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540
Dates: Start 2001-07; Study Completion 2002-07

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation for Fighting Blindness, Baltimore, Maryland, United States